CLINICAL TRIAL: NCT02037022
Title: Pivotal Response Treatment Package for Young Children With Autism
Acronym: PRT-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-28314; R21DC013689 (NIH)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder (ASD); Autism
Keywords: Autism Spectrum Disorder (ASD); Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pivotal Response Treatment Package (Experimental): Pivotal Response Treatment Package (PRT-P)
  Interventions: Behavioral: Pivotal Response Treatment Package (PRT-P)
- Delayed Treatment Group (No Intervention): Delayed Treatment Group (DTG)

INTERVENTIONS:
Behavioral: Pivotal Response Treatment Package (PRT-P)
  Arms: Pivotal Response Treatment Package

SUMMARY:
This is a research study examining the effectiveness of a pivotal response treatment package (PRT-P) in targeting language skills in young children with autism.

DETAILED DESCRIPTION:
Researchers at the Stanford University School of Medicine are seeking participants for a research study examining the effectiveness of a pivotal response treatment package (PRT-P) in targeting language skills in young children with autism. Research has demonstrated that behavioral interventions, such as Pivotal Response Training (PRT), lead to improvements in the core symptoms of autism. Researchers have begun to develop strategies to investigate the effectiveness of combining a parent training program teaching parents how to implement PRT with in-home, therapist-implemented treatment. To determine the effectiveness of a PRT-P, it will be compared to a delayed treatment group (DTG) by conducting a randomized controlled 24-week trial. This research will allow us to help in the development of therapeutic approaches that can meet the increasing service demands for families. We hope that investigating interventions that aim to improve core deficits will aid clinicians in providing better care for children with autism.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) based on Autism Diagnostic Interview- Revised (ADI-R), Autism Diagnostic Observation Schedule (ADOS-2), and expert clinical opinion
* Males and females in good medical health between 2.0 and 5.11 years
* Ability to participate in the testing procedures to the extent that valid standard scores can be obtained
* Language delay as measured by the Preschool Language Scale: Standard score at least 1 Standard Deviation below average for expressive language ability
* Stable treatment, speech therapy, school placement, psychotropic medication(s) or biomedical intervention(s) for at least 1 month prior to baseline measurements with no anticipated changes during study participation
* No more than 60 minutes of individual 1:1 speech therapy per week
* Availability of at least one parent who can consistently participate in parent training and research measures
* Parents intend on continuing Pivotal Response Treatment Package (PRT-P) for a minimum of 12 weeks
* Parents must be 18 years of age or older

Exclusion Criteria:

* Current or lifetime diagnosis of severe psychiatric disorder, such as bipolar disorder
* Receiving in-home Applied Behavior Analysis (ABA) of 10 hours or more
* A genetic abnormality, such as Fragile X
* Presence of active medical problem, such as unstable seizure disorder or heart disease
* Previous adequate PRT trial
* Participants living more than 50 miles from Stanford University
* At least one room of the house must be available to be dedicated to treatment during session times
* There must be no serious health and safety risks present in the home environment
* The research team has the right to refuse to perform sessions in-home even if the criteria above are met

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2013-12-04 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in communication during parent-child and clinician-child interactions at 6, 12, and 24 weeks | 6, 12 and 24 weeks

SECONDARY OUTCOMES:
Change from Baseline on the Preschool Language Scale, 5th Edition (PLS-5) at 12, and 24 weeks | 12 and 24 weeks
Change from Baseline on the Sensory Profile Questionnaire at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline on the Social Responsiveness Scale (SRS) at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline on the MacArthur-Bates Communication Development Inventory at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline on the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline on the Behavior Rating Inventory of Executive Function, Preschool (BRIEF-P) at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline on the Parenting Stress Index (PSI) at 6, 12, and 24 weeks | 6, 12, and 24 weeks
Change from Baseline on the Family Empowerment Scale (FES) at 6, 12, and 24 weeks | 6, 12, and 24 weeks
Change from Baseline on the Clinical Global Impression Scale at 6, 12, and 24 weeks | 6, 12, and 24 weeks
Change from Baseline on the Social attention and word-learning eye tracking task at 12, and 24 weeks | 12, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Gengoux GW, Abrams DA, Schuck R, Millan ME, Libove R, Ardel CM, Phillips JM, Fox M, Frazier TW, Hardan AY. A Pivotal Response Treatment Package for Children With Autism Spectrum Disorder: An RCT. Pediatrics. 2019 Sep;144(3):e20190178. doi: 10.1542/peds.2019-0178. Epub 2019 Aug 6. PMID 31387868
- [Derived] Gengoux GW, Schapp S, Burton S, Ardel CM, Libove RA, Baldi G, Berquist KL, Phillips JM, Hardan AY. Effects of a parent-implemented Developmental Reciprocity Treatment Program for children with autism spectrum disorder. Autism. 2019 Apr;23(3):713-725. doi: 10.1177/1362361318775538. Epub 2018 May 18. PMID 29775078